CLINICAL TRIAL: NCT06486441
Title: A Randomized, Open-label, Phase 3 Study of Sacituzumab Govitecan Versus Treatment of Physician's Choice in Participants With Endometrial Cancer Who Have Received Prior Platinum-based Chemotherapy and Anti-PD-1/PD-L1 Immunotherapy
Brief Title: Study of Sacituzumab Govitecan Versus Treatment of Physician's Choice in Participants With Endometrial Cancer After Platinum-Based Chemotherapy and Immunotherapy (ASCENT-GYN-01/GOG-3104/ENGOT-en26)
Acronym: ASCENT-GYN-01
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: GOG Foundation (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Asia-Pacific Gynecologic Oncology Trials Group (APGOT) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-682-6769; 2024-511957-23 (Other: European Medicines Agency); GOG-3104 (Other: The GOG Foundation); ENGOT-en26 (Other: European Network for Gynaecological Oncological Trial Groups); APGOT-EN2 (Other: Asia-Pacific Gynecologic Oncology Trials Group)
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — sacituzumab govitecan; Doxorubicin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sacituzumab Govitecan (SG) (Experimental): Participants will receive SG at a dose of 10 mg/kg on Days 1 and 8 of a 21-day cycle.
  Interventions: Drug: Sacituzumab govitecan-hziy
- Treatment of Physician's Choice (TPC) (Active Comparator): Participants will receive one of the following TPC, regimens determined prior to randomization.
  * Doxorubicin 60 mg/m^2 IV on Day 1 of a 21-day cycle
  * Paclitaxel 80 mg/m^2 IV on Days 1, 8, and 15 of a 28-day cycle
  Interventions: Drug: Doxorubicin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Sacituzumab govitecan-hziy — Administered intravenously
  Other Names: Trodelvy™; GS-0132
  Arms: Sacituzumab Govitecan (SG)
Drug: Doxorubicin — Administered intravenously
  Other Names: Adriamycin
  Arms: Treatment of Physician's Choice (TPC)
Drug: Paclitaxel — Administered intravenously
  Other Names: Taxol
  Arms: Treatment of Physician's Choice (TPC)

SUMMARY:
The goal of this clinical study is to find out how the study drug, sacituzumab govitecan (SG) works in participants with endometrial cancer who have received prior treatment with platinum-based chemotherapy and immunotherapy, versus the treatment of physician's choice (TPC).

The primary objectives of this study are to evaluate the effect of SG compared to TPC on progression-free survival (PFS) as assessed by blinded independent central review (BICR) and overall survival (OS).

ELIGIBILITY:
Key Inclusion Criteria:

* Documented evidence of recurrent/persistent endometrial cancer (endometrial carcinoma or carcinosarcoma).
* Up to 3 prior lines of systemic therapy for endometrial cancer, including systemic platinum-based chemotherapy and anti-PD-1/PD-L1 therapy, either in combination or separately.
* Eligible for treatment with either doxorubicin or paclitaxel as determined by the investigator.
* Radiologically evaluable disease (either measurable or nonmeasurable) by computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST v1.1.
* Eastern Cooperative Oncology Group performance status score of 0 or 1.
* Adequate organ function

Key Exclusion Criteria:

* Uterine leiomyosarcoma and endometrial stromal sarcomas are excluded.
* Participants who are candidates for curative-intent therapy at the time of study enrollment.
* Participants eligible for rechallenge with platinum-based chemotherapy as determined by the investigator.
* Received any prior treatment with a Trop-2-directed antibody-drug conjugate (ADC).
* Have an active second malignancy.
* Have an active serious infection requiring systemic antimicrobial therapy.
* Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or gastrointestinal perforation within 6 months prior to randomization.
* Have a positive serum pregnancy test or are breastfeeding for participants who are assigned female at birth.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 640 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) As Assessed by Blinded Independent Central Review (BICR) | Up to approximately 27 months
  PFS, defined as the time from the date of randomization until the date of objective progressive disease (PD), as assessed by BICR per Response Evaluation Criteria in Solid Tumors (RECIST v1.1), or death from any cause, whichever comes first.
Overall Survival (OS) | Up to approximately 47 months
  Overall survival (OS) is defined as time from the date of randomization until death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by BICR | Up to approximately 47 months
  ORR, defined as the percentage of participants who have achieved a CR or PR as best overall response that is confirmed ≥ 4 weeks after initial documentation of response as assessed by BICR per RECIST v1.1.
Change from Baseline in the Physical Functioning Domain of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 Version 3.0 (EORTC QLQ-C30) at Week 16 | Baseline, Week 16
  The EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients, it is composed of 30 questions (items) resulting in 5 functional scales, 1 global health status scale, 3 symptom scales, and 6 single items. Scoring of the QLQ-C30 is performed according to QLQ-C30 Scoring manual. The physical functioning scale range in score from 0 to 100. Higher score denote a better level of functioning (i.e. a better state of the participant).
PFS as Assessed by Investigator | Up to approximately 27 months
  PFS is defined as the time from the date of randomization until the date of objective PD, as assessed by investigator per RECIST v1.1, or death from any cause, whichever comes first
ORR as Assessed by Investigator | Up to approximately 47 months
  ORR is defined as the percentage of participants who have achieved a CR or PR as best overall response that is confirmed ≥ 4 weeks after initial documentation of response as assessed by investigator per RECIST v1.1
Duration of Response (DOR) as Assessed by BICR and Investigator | Up to approximately 47 months
  DOR is defined as the time from the first documentation of CR or PR to the earlier of the first documentation of definitive PD as assessed by BICR and investigator per RECIST v1.1, or death from any cause, whichever comes first.
Clinical Benefit Rate (CBR) as Assessed by BICR and Investigator | Up to approximately 47 months
  CBR is defined as the percentage of participants with best overall response of CR or PR that is confirmed ≥ 4 weeks after initial documentation of response or durable stable disease (SD; duration of SD ≥ 6 months from randomization to disease progression), as assessed by BICR and investigator per RECIST v1.1.
Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs) | First dose date up to 30 days post last dose (Up to Up to approximately 47 months)
Percentage of Participants Experiencing Clinical Laboratory Abnormalities | First dose date up to 30 days post last dose (Up to Up to approximately 47 months)
Change from baseline in Global Health Status (GHS)/Quality of Life (QoL) Domain of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 Version 3.0 (EORTC QLQ-C30) at Week 16 | Baseline, Week 16
  The EORTC QLQ-C30 is a questionnaire to assess quality of life of cancer patients, it is composed of 30 questions (items) resulting in 5 functional scales, 1 global health status scale, 3 symptom scales, and 6 single items. Scoring of the QLQ-C30 is performed according to QLQ-C30 Scoring manual. Global health status score ranges from 0 to 100. Higher score denote a better level of functioning (i.e. a better state of the participant).

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (189):
- United States (57):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - UC San Diego Medical Center, La Jolla, California
  - Cedars-Sinai Cancer at Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford Women's Cancer Center, Palo Alto, California
  - Kaiser Permanente Medical Center, Vallejo, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - Hartford HealthCare Cancer Institute at Hartford Hospital, Hartford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Florida Cancer Specialists, Fort Myers, Florida
  - University of Florida, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Lewis Cancer & Research Pavilion at St. Joseph's/Candler Health System, Savannah, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - M Health Fairview University of Minnesota Medical Center - East Bank Hospital, Minneapolis, Minnesota
  - Metro Minnesota Community Oncology Research Consortium (MMCORC), Saint Louis Park, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - MidAmerica Division, Inc. c/o Research Medical Center, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health Cancer Institute, Lake Success, New York
  - Columbia University Medical Center, Herbert Irving Pavilion, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Oklahoma Cancer Specialists and Research Institute - OCSRI - Tulsa, Tulsa, Oklahoma
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Alliance Cancer Specialists, PC, Horsham, Pennsylvania
  - University of Pennsylvania Health System, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - SCRI Oncology Partners, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology, Fort Worth, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Froedtert and the Medical College of Wisconsin (MCW), Milwaukee, Wisconsin
- Australia (6):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Mater Cancer Care Centre, South Brisbane, Queensland
  - Monash Health, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Murdoch, Western Australia
- Brazil (9):
  - Clínica de Neoplasias Litoral, Itajaí
  - Centro de Pesquisa Clínica do Hospital Moinhos de Vento, Porto Alegre
  - Hospital Santa Joana Recife, Recife
  - Instituto D'Or Pesquisa e Ensino, Rio de Janeiro
  - Ensino e Terapia de Inovação Clínica AMO - ETICA, Salvador
  - Instituto do Câncer do Estado de São Paulo, São Paulo
  - BP - A Beneficência Portuguesa da São Paulo / Hospital BP Mirante, São Paulo
  - DASA - Hospital 9 de Julho, São Paulo
  - AC Camargo Cancer Center (Fundação Antonio Prudente), São Paulo
- Canada (6):
  - Arthur J. E. Child Comprehensive Cancer Centre, Calgary
  - London Health Sciences Centre, London
  - McGill University Health Centre - Glen Site, Montreal
  - CIC-CHU de Québec-Université Laval- Hôpital de l'Enfant-Jésus, Québec
  - Sunnybrook Research Institute, Toronto
  - Princess Margaret Cancer Centre, Toronto
- China (18):
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Second Hospital of Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Guangxi Medical University Affiliated Tumor Hospital, Guangxi Zhuang Autonomous Region
  - Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou
  - Women's Hospital School Of Medicine Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Jiangxi Maternal and Child Health Hospital, Nanchang
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou
- Czechia (4):
  - Nemocnice AGEL, Nový Jičín a.s., Nový Jičín
  - University Hospital Ostrava, Ostrava-Poruba
  - General University Hospital in Prague, Prague
  - University Hospital Bulovka, Prague
- France (8):
  - Centre Francois Baclesse, Caen
  - Institut Paoli Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Hôpital Cochin, Paris
  - HCL - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - ICO - Centre René Gauducheau, Saint-Herblain
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (8):
  - Hochtaunus Kliniken Bad Homburg, Bad Homburg
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - University Hospital Essen, Essen
  - Universitätsklinikum Hamburg, Hamburg
  - Medical School Hannover, Hanover
  - University Hospital Leipzig, Leipzig
  - Klinikum rechts der Isar der TU München, Klinik und Poliklinik für Frauenheilkunde, München
  - Universitätsklinikum Ulm, Ulm
- Greece (5):
  - Aretaeion Hospital, Athens
  - MITERA hospital, Athens
  - Kalamata Hospital, Kalamata
  - General Hospital of Patras Agios Andreas, Pátrai
  - St. Luke's Hospital, Thessaloniki
- Hong Kong (3):
  - Hong Kong Sanatorium & Hospital, Happy Valley
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, New Territories
- Israel (6):
  - Hillel Yaffe Medical Center, Hadera
  - Rambam Health Care Campus, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Sourasky T.A.M.C., Tel Aviv
- Italy (13):
  - SOC di Oncologia Medica e Prevenzione Oncologica Centro di Riferimento Oncologico di Aviano (CRO) IRCCS, Aviano
  - Azienda Ospedaliera Universitaria Careggi - Unita di Oncologia Ginecologica, Florence
  - ASST Lecco - Ospedale Alessandro Manzoni, Lecco
  - Istituto Romagnolo per lo Studio dei Tumori-Dino Amadori - IRST, Meldola
  - Irccs Ospedale San Raffaele-UO Ginecologia, Milan
  - Fondazione IRCCS - Istituto Nazionale dei Tumori di Milano, Milan
  - Istituto Europeo di Oncologia, Milan
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero Universitaria Pisana, Ospedale Santa Chiara, Pisa
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Istituto Nazionale Tumori Regina Elena IRCCS, Rome
  - AOU Città della Salute e della Scienza di Torino - Presidio Sant'Anna, Torino
  - A.O. Ordine Mauriziano di Torino, Torino
- Japan (10):
  - Chiba Cancer Center, Chiba
  - The Jikei University Kashiwa Hospital, Chiba
  - Hyogo Cancer Center, Hyōgo
  - St. Marianna University Hospital, Kanagawa
  - Mie University Hospital, Mie
  - Okayama University Hospital, Okayama
  - Saitama Medical University International Medical Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital Of JFCR, Tokyo
- Poland (5):
  - Szpitale Pomorskie Sp. z o.o., Gdynia
  - Uniwersyteckie Centrum Kliniczne SUM, Katowice
  - Oddział Ginekologii Onkologicznej Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Mazowiecki Szpital Wojewódzki im. św. Jana Pawła II w Siedlcach, Siedlce
  - Dolnoslaskie Centrum Onkologii, Wroclaw
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (6):
  - Keimyung University Dongsan Medical Center, Dalseo-gu
  - National Cancer Center - Korea, Goyang-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Seoul
- Spain (11):
  - Complexo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Ciudad de Jaen, Jaén
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitari Son Espases, Palma
  - Hospital Parc Taulí, Sabadell
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitario La Fe - Valencia, Valencia
- Taiwan (6):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- United Kingdom (6):
  - Birmingham Heartlands Hospital, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - University Hospitals of Leicester NHS Trust-Leicester Royal Infirmary, Leicester
  - University College London Hospitals, London
  - East and North Hertfordshire NHS Trust - Mount Vernon Cancer Centre, Northwood

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eskander RN, Corr B, Cibula D, Tan DSP, Cloven N, Guerra E, Hasegawa K, Myers T, You B, Makker V, Zagouri F, Gien LT, Bartoletti M, Mallen A, Woelber L, Mocci S, Komatsubara K, Ma L, Colombo N. A randomized, phase III study of sacituzumab govitecan versus treatment of the physician's choice in patients with endometrial cancer after platinum-based chemotherapy and immunotherapy: the ASCENT-GYN-01 study (GOG-3104/ENGOT-en26/APGOT-EN2). Int J Gynecol Cancer. 2025 Sep 7:102654. doi: 10.1016/j.ijgc.2025.102654. Online ahead of print. PMID 41073155
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06486441